CLINICAL TRIAL: NCT04998565
Title: Comparing the add-on Effectiveness of Electro-acupuncture or Transcutaneous Electrical Nerve Stimulation in Early Postpartum Breast Engorgement: A Pilot Randomized Pragmatic Trial
Brief Title: Add-on Effectiveness of EA or TENS in Early Postpartum Breast Engorgement
Acronym: ETBEG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No grants from the Ministry of Science and Technology or school grants, no funds can be executed, so the application is terminated.
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH106-REC1-101
Record Dates: First submitted 2017-10-08; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Breast Engorgement in Puerperium; Post Partum Depression
Keywords: Electrical acupuncture; Transcutaneous Electrical Nerve Stimulation
MeSH Terms: conditions — Depression, Postpartum | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine care (Experimental): Routine care for early postpartum breast engorgement, including reverse pressure technique over areola, along with hand expression of breastmilk.
  Interventions: Other: Routine care
- Routine care plus EA (Experimental): Routine care for early postpartum breast engorgement, including reverse pressure technique over areola, along with hand expression of breastmilk.
  plus: Electrical acupuncture on body acupoints
  Interventions: Other: Routine care; Procedure: Electrical Acupuncture
- Routine care plus TENS (Experimental): Routine care for early postpartum breast engorgement, including reverse pressure technique over areola, along with hand expression of breastmilk.
  plus: Transcutaneous electrical nerve stimulation on breasts
  Interventions: Other: Routine care; Procedure: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Other: Routine care — Reverse pressure applied to the areola
Procedure: Electrical Acupuncture — Acupuncture on Hegu, Sanyinjiao, Zusanli and Taichong with electrical stimulation
  Arms: Routine care plus EA
Procedure: Transcutaneous Electrical Nerve Stimulation — Transcutaneous electrical nerve stimulation over bil breasts
  Arms: Routine care plus TENS

SUMMARY:
A total of 36 volunteers of postpartum women within 7 days with significant breast engorgement, will be recruited in China Medical University Hospital, Taichung, Taiwan. The participants will be randomly assigned into 3 groups, each of 12 people, namely, routine care group, routine care plus electrical-acupuncture experiment group, and routine care plus transcutaneous electrical nerve stimulation group.

DETAILED DESCRIPTION:
Participants will receive once a day, three consecutive days of interventions in each group, including identical routine care. On each visit, severity index (SI) subject to the extent of erythema, tension and pain over breast will be assessed. Questionnaires of Breastfeeding Self-Efficacy Scale (BSES-SF) and of Edinburgh postnatal depression scale (EPDS) will be performed. Heart-rate variability was evaluated and recorded via a real-time handheld HRV device. Oxycontin, Cortisol, sodium and potassium levels in breastmilk will be tested . A telephone follow-up will be performed in 30 days after completion of treatment, and the data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 37 wk
* Delivery of singleton, healthy newborn baby
* Within 7 days postpartum
* Within 24 hours from initial painful breast engorgement
* Difficulty on lactation due to plugged ducts, SI index ≧ 5 (0-19)

Exclusion Criteria:

* Fever>37.5∘C
* Mastitis or breast abscess
* Signs of sepsis or other infection
* Perinatal mother and infant diseases (Gestational hypertension、Gestational Diabetes Mellitus、Pre-eclampsia 、Gestational thyroid diseases or Intrauterine growth retardation)
* Psychological diseases
* Bleeding tendency
* Artificial valves
* Pacemaker
* Epilepsy
* Consciousness disturbance
* Skin infections
* Hepatitis B carrier
* Acquired Immune Deficiency Syndrome
* Breast tumors
* Breast Surgeries

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Postpartum women
Enrollment: 2 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Severity Index (0-19) | Changes from Baselines of Severity Index, at each treatment and 1 month later
  Sum of the degree of Erythema, Tension and Pain scores over breasts

SECONDARY OUTCOMES:
EPDS | Changes from Baseline of EPDS, after each treatment and 1 month later
  Edinburgh Postnatal Depression Scale
BSES-SF | Changes from Baseline of BEES-SF, after each treatment and 1 month later
  Breastfeeding Self-Efficacy Scale

OTHER OUTCOMES:
HRV | Change from Baseline of HRV, immediately after each treatment
  Real-time handheld Heart-rate Variability
Lab Data | Changes from Baseline of Oxytocin and Cortisol levels, immediately after each treatment
  Measurements of Oxytocin and Cortisol levels in breastmilk

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Rong Yen, PhD, Study Chair — Department of Chinese Medicine, China Medical University
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No